CLINICAL TRIAL: NCT06256640
Title: Mandibular Advancement Device (MAD) as an Alternative Treatment Option in Pregnant Women With Obstructive Sleep Apnea (OSA)
Brief Title: Mandibular Advancement Device (MAD) in Pregnant Women With Obstructive Sleep Apnea (OSA)
Acronym: OBMAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll participants
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15984-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea of Adult; Pregnancy Related
MeSH Terms: interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: Mandibular advancement Device

INTERVENTIONS:
Device: Mandibular advancement Device — Intra oral appliances and more specifically Mandibular Advance Devices (MAD) are one of the established alternatives to treat OSA. Oral appliances and MAD are often used interchangeably but we prefer to call them MAD as it is more descriptive of its mechanism of action. MAD are placed in the mouth to temporarily advance and stabilize the lower jaw forward in order to keep the airway open during sleep.

SUMMARY:
We propose a single-arm trial to test the patient uptake and preliminary efficacy of MAD in a sample of 10 pregnant women with mild-to-moderate OSA. Study outcomes include patient-reported symptoms and objectively assessed sleep parameters assessed before treatment, during and after 10 weeks of MAD intervention (during pregnancy) and postpartum.

DETAILED DESCRIPTION:
The purpose of this study is to explore MAD as an alternative treatment option for OSA in pregnant women. We are recruiting a small number of 10 healthy pregnant women with uncomplicated OSA (absence of significant cardiovascular, metabolic or neurocognitive consequences) who, after being offered CPAP as the recommended standard treatment, prefer to use a MAD over CPAP. All patients are recruited from a single center. We would like to get a first impression on the comfort level of these women with the MAD and their self-reported compliance and any improvement of symptoms with treatment. Additionally, we would like to test efficacy in controlling OSA with pregnancy progression. Finally, we would like to derive overall treatment effectiveness of the MAD in pregnant women as defined as a combination of efficacy and compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy, gestational week 14-20.
2. Age ≥ 18, English-speaking.
3. Reliable internet access (questionnaires/surveys)
4. Untreated mild to mild-moderate OSA defined as AHI between 5-20 events/hour on the most recent home sleep study
5. No significant hypoxemia on the initial sleep study defined as SaO2 nadir ≥70% and SaO2 equal or less than 30 minutes ≥88%
6. The sleep study must have been a home sleep test that uses Peripheral Arterial Tone signal for evaluation of apneic events. The home sleep test has to be a WatchPAT device (WatchPAT® Home Sleep Study Device | Itamar Medical Ltd.).
7. No significant confounding comorbidities including restless leg symptoms and circadian disorders (shift work)
8. BMI less or equal to 40 and neck size less or equal to 40 cm
9. Good oral health with manual dexterity and at least 8 tooth per arch

Exclusion Criteria:

1. High risk pregnancy (age >40y, superimposed preeclampsia, pre-existing cardiac disease, severe organ dysfunction such as liver or renal failure, any condition that requires anticoagulation), and any condition Dr. Pitts or Dr Smith deem serious risk to mother/fetus. Well controlled chronic hypertension and diabetes are allowed and will not be excluded.
2. Dental exclusion criteria: Complete edentulous arch, ongoing oral rehabilitation, uncontrolled periodontal disease, ongoing orthodontic treatment or completed treatment in a period less than 5 years, temporomandibular dysfunction (active acute pain or limitations on mandibula movements of any kind), prior oropharyngeal surgery, maximum protrusion less 5 mm
3. Significant acute health problems that are unrelated to pregnancy or dental diseases including unstable psychiatric disease
4. Non-English speaking
5. Unable to provide informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 0 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Describe patient uptake of MAD | 9 months
  MAD adherence will be determined via patient-reported sleep diaries during the first 10-weeks of MAD intervention according to the AADSM guidelines. Specifically, patients will report each morning whether they wore their MAD and to estimate how long they wore it for. Consistent with Medicare guidelines for PAP therapy, we will operationalize compliance as wearing the device for ≥4 hrs each night for 70% of nights. We will describe compliance rates.
Evaluate preliminary efficacy of MAD for treating mild-to-moderate OSA | 9 months
  We will assess AHI before treatment (T1), after 10 weeks of MAD treatment during pregnancy (T2), and then finally three months after childbirth (T3) via home sleep tests used in our sleep clinic per standard care. We hypothesize that AHI at T2 and T3 will be significantly lower than T1. For descriptive purposes, we will report rates of OSA remission (AHI<5) at T2 and T3 as well as rates of positive treatment response operationalized as a ≥50% reduction in AHI from T1.
Test for changes in patient-reported symptoms. | 9 months
  OSA is associated with increased fatigue and sleepiness. We hypothesize that patients will report lower levels of fatigue and daytime sleepiness at T2 and T3 relative to T1 baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Jaziri, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided